CLINICAL TRIAL: NCT00461851
Title: A Phase II, Multicenter Trial of Gemcitabine, Carboplatin, and Sorafenib in Chemotherapy-naive Patients With Advanced/Metastatic Bladder Carcinoma
Brief Title: Trial of Gemcitabine, Carboplatin, and Sorafenib in Chemotherapy-naive Patients With Advanced/Metastatic Bladder Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0609001823
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2016-09

CONDITIONS: Bladder Cancer
Keywords: Advanced/Metastatic Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Carboplatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy plus sorafenib (Experimental): Gemcitabine 1000 mg/m2 weekly x 2 weeks plus carboplatin AUC (Area under curve) 5 every 3 weeks plus sorafenib x 6 cycles then maintenance sorafenib alone
  Interventions: Drug: Gemcitabine; Drug: Carboplatin; Drug: Sorafenib

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be given at a standard dose schedule of 1000 mg/m² on day 1 and 8.
  Other Names: Gemzar
Drug: Carboplatin — Carboplatin will be given on day 1 to an AUC of 5.
Drug: Sorafenib — Sorafenib will be administered orally daily on days 2-19 at 400 mg bid
  Other Names: BAY 43-9006

SUMMARY:
This is a Phase II, nonrandomized multicenter study designed to evaluate time to progression and response proportion of patients with advanced or metastatic transitional cell carcinoma of bladder receiving 6 cycles of gemcitabine, carboplatin and sorafenib and then maintenance sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of diagnosis of transitional cell carcinoma of the bladder, urethra, ureter, or renal pelvis
* Unresectable, locally advanced or metastatic disease
* CrCl ≥ 60 ml/min or serum creatinine < 1.5
* ≥ 4 weeks since prior RT
* ECOG Performance Status of 0 or 1 (Appendix I)
* Age ≥ 18 years of age
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men and women should use adequate birth control for at least 2 weeks after the last administration of sorafenib.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin > 9.0 g/dl
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Total bilirubin ≤ 1.5 times ULN
* ALT and AST ≤ 2.5 times the ULN ( ≤ 5 x ULN for patients with liver involvement)
* INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.

Exclusion Criteria:

* Prior treatment with systemic chemotherapy (prior intravesical chemotherapy is permitted, and adjuvant therapy is permitted if > 12 months have lapsed)
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study
* Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* History of stroke within six months
* Clinically significant peripheral vascular disease
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Sorafenib is contraindicated in patients with known severe hypersensitivity to sorafenib or any of the excipients.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > CTCAE Grade 2.
* Thrombolytic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, significant traumatic injury within 4 weeks of first study drug
* Use of St. John's Wort or rifampin (rifampicin)
* Known or suspected allergy to sorafenib or any agent given in the course of this trial
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem
* Anticipation of need for major surgical procedure during the course of the study
* Pregnant (positive pregnancy test) or lactating
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures
* History of persistent gross hematuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hari Deshpande, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, Comprehensive Cancer Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 19 patients were screened, 17 enrolled in the study.
Period: Overall Study
Arm/Group | Chemotherapy Plus Sorafenib
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy Plus Sorafenib
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 65 [47 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The primary outcome was the proportion of patients who achieved progression free survival (PFS) of five months. PFS was defined as time to progression or any-cause mortality, whichever came first.
Time Frame: Upon completion of study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Plus Sorafenib
Number analyzed (Participants) | 17
months | 9.5 [5.6 to 16.4]

2. Secondary Outcome: Dose Ruction (Toxicity)
Description: To determine the toxicity of combination therapy with sorafenib, gemcitabine and carboplatin, dose reductions by drug are reported. The number of patients that were reduced in dosage are reported here.
Time Frame: Upon completion of study
Population: 17 patients were evaluable for toxicity. A total of 77 cycles of gemcitabine/carboplatin were administered with a median 4.5 cycles per patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Plus Sorafenib
Number analyzed (Participants) | 17
Participants
  Dose Reduction: Gemcitabine | 15
  Dose Reduction: Carboplatin | 5
  Dose Reduction: Sorafenib | 9

3. Secondary Outcome: Best Reported Response
Description: The best reported response captures the proportion of patients with advanced or metastatic transitional cell carcinoma of the bladder that achieve a complete or partial response to the combination therapy with sorafenib, gemcitabine, and carboplatin.
Time Frame: Upon completion of study
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Plus Sorafenib
Number analyzed (Participants) | 17
Participants
  Partial Response | 5
  Complete Response | 4
  Stable Disease | 7
  Lost to Follow Up | 1

ADVERSE EVENTS:
Arm/Group | Chemotherapy Plus Sorafenib
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Plus Sorafenib (N=17)
Hospitalization for sepsis (Infections and infestations) | 1 (1)
MI (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No